CLINICAL TRIAL: NCT02312154
Title: Split-face Study of Changing in Skin Physiology and Clinical Appearance After Microdroplet Placement of Stabilized Hyaluronic Acid in Aging Faces
Brief Title: Changing in Skin Physiology After Microdroplet Placement of Stabilized Hyaluronic Acid in Aging Faces
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Konkuk University Hospital (Other)
Responsible Party: Principal Investigator, Yang Won Lee, Professor, Konkuk University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: KUH1120048
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Results first posted 2015-02-24 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Aging

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treated side (Restylane vital) (Experimental): We injected staabilized hyaluronic acid (HA)-based gel of nonanimal origin on the left side of face.
  (We performed split face study)
  Interventions: Device: Restylane Vital
- untreated side (control) (No Intervention): We did nothing on the right side of face and we compared the results on same participants

INTERVENTIONS:
Device: Restylane Vital — stabilized hyaluronic acid (HA)-based gel of nonanimal origin
  Arms: treated side (Restylane vital)

SUMMARY:
IMPORTANCE Skin rejuvenation can be achieved effectively and safely by injection of a stabilized hyaluronic acid (HA)-based gel of nonanimal origin (NASHA) injection using a stamp-type electronic multineedle injector.

OBJECTIVE To determine the efficacy and safety of NASHA using a stamp-type electronic multineedle injector, and if changes in skin physiology occur earlier than in previous trials.

DESIGN, SETTING, AND PARTICIPANTS Twenty-five patients were recruited to this single-center, evaluator-blinded, prospective, balanced (1:1), split-face randomized clinical trial.One dermatologist who was blinded as to the treatment side evaluated the skin hydration, melanin content, erythema, and elasticity of both cheeks using a corneometer, a mexameter, and a reviscometer, respectively, at each follow-up visit (0, 1, 2, 4, 8, and 12 weeks postinjection). The subjects and two independent investigators assessed the clinical improvement using the Global Aesthetic Improvement Scale (GAIS) at the every visit. Twenty-four participants completed the study, and no participants withdrew due to adverse effects.

INTERVENTIONS Each participant submitted to a single treatment with a NASHA injection to one side of the lower cheek. The cheek side to which the treatment was applied was chosen randomly.

DETAILED DESCRIPTION:
Twenty-five patients were recruited to this single-center, evaluator-blinded, prospective, balanced (1:1), split-face randomized clinical trial. Twenty-four participants completed the study, and no participants withdrew due to adverse effects. Each participant submitted to a single treatment with a NASHA injection to one side of the lower cheek. One dermatologist who was blinded as to the treatment side evaluated the skin hydration, melanin content, erythema, and elasticity of both cheeks using a corneometer, a mexameter, and a reviscometer, respectively, at each follow-up visit (0, 1, 2, 4, 8, and 12 weeks postinjection). The subjects and two independent investigators assessed the clinical improvement using the Global Aesthetic Improvement Scale (GAIS) at the every visit. Adverse events were self-reported by the patients completing a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Healthy people older than 25 years

Exclusion Criteria:

* known hypersensitivity to HA, an active skin disease, any autoimmune disorder, or significant renal, hepatic, or other medical diseases

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yang Won Lee, MD, PhD, Principal Investigator — Department of Dermatology, Konkuk University School of Medicine, Seoul, Korea

REFERENCES:
- [Background] Gniadecka M, Nielsen OF, Wessel S, Heidenheim M, Christensen DH, Wulf HC. Water and protein structure in photoaged and chronically aged skin. J Invest Dermatol. 1998 Dec;111(6):1129-33. doi: 10.1046/j.1523-1747.1998.00430.x. PMID 9856828
- [Background] Matarasso SL, Carruthers JD, Jewell ML; Restylane Consensus Group. Consensus recommendations for soft-tissue augmentation with nonanimal stabilized hyaluronic acid (Restylane). Plast Reconstr Surg. 2006 Mar;117(3 Suppl):3S-34S. doi: 10.1097/01.prs.0000204759.76865.39. PMID 16531934
- [Background] Kerscher M, Bayrhammer J, Reuther T. Rejuvenating influence of a stabilized hyaluronic acid-based gel of nonanimal origin on facial skin aging. Dermatol Surg. 2008 May;34(5):720-6. doi: 10.1111/j.1524-4725.2008.34176.x. Epub 2008 Apr 1. PMID 18384619
- [Background] Streker M, Reuther T, Krueger N, Kerscher M. Stabilized hyaluronic acid-based gel of non-animal origin for skin rejuvenation: face, hand, and decolletage. J Drugs Dermatol. 2013 Sep;12(9):990-4. PMID 24002145
- [Background] Naylor EC, Watson RE, Sherratt MJ. Molecular aspects of skin ageing. Maturitas. 2011 Jul;69(3):249-56. doi: 10.1016/j.maturitas.2011.04.011. Epub 2011 May 25. PMID 21612880
- [Background] Distante F, Pagani V, Bonfigli A. Stabilized hyaluronic acid of non-animal origin for rejuvenating the skin of the upper arm. Dermatol Surg. 2009 Feb;35 Suppl 1:389-93; discussion 394. doi: 10.1111/j.1524-4725.2008.01051.x. No abstract available. PMID 19207331
- [Background] Williams S, Tamburic S, Stensvik H, Weber M. Changes in skin physiology and clinical appearance after microdroplet placement of hyaluronic acid in aging hands. J Cosmet Dermatol. 2009 Sep;8(3):216-25. doi: 10.1111/j.1473-2165.2009.00447.x. PMID 19735521
- [Background] Reuther T, Bayrhammer J, Kerscher M. Effects of a three-session skin rejuvenation treatment using stabilized hyaluronic acid-based gel of non-animal origin on skin elasticity: a pilot study. Arch Dermatol Res. 2010 Jan;302(1):37-45. doi: 10.1007/s00403-009-0988-9. PMID 19730872
- [Background] Ribe A, Ribe N. Neck skin rejuvenation: histological and clinical changes after combined therapy with a fractional non-ablative laser and stabilized hyaluronic acid-based gel of non-animal origin. J Cosmet Laser Ther. 2011 Aug;13(4):154-61. doi: 10.3109/14764172.2011.594060. Epub 2011 Jun 23. PMID 21699363
- [Background] Tezel A, Fredrickson GH. The science of hyaluronic acid dermal fillers. J Cosmet Laser Ther. 2008 Mar;10(1):35-42. doi: 10.1080/14764170701774901. PMID 18330796
- [Background] Wang F, Garza LA, Kang S, Varani J, Orringer JS, Fisher GJ, Voorhees JJ. In vivo stimulation of de novo collagen production caused by cross-linked hyaluronic acid dermal filler injections in photodamaged human skin. Arch Dermatol. 2007 Feb;143(2):155-63. doi: 10.1001/archderm.143.2.155. PMID 17309996
- [Background] Alam M, Han S, Pongprutthipan M, Disphanurat W, Kakar R, Nodzenski M, Pace N, Kim N, Yoo S, Veledar E, Poon E, West DP. Efficacy of a needling device for the treatment of acne scars: a randomized clinical trial. JAMA Dermatol. 2014 Aug;150(8):844-9. doi: 10.1001/jamadermatol.2013.8687. PMID 24919799
- [Background] Kim SE, Lee JH, Kwon HB, Ahn BJ, Lee AY. Greater collagen deposition with the microneedle therapy system than with intense pulsed light. Dermatol Surg. 2011 Mar;37(3):336-41. doi: 10.1111/j.1524-4725.2011.01882.x. Epub 2011 Feb 22. PMID 21342311
- [Background] Lim HK, Suh DH, Lee SJ, Shin MK. Rejuvenation effects of hyaluronic acid injection on nasojugal groove: prospective randomized split face clinical controlled study. J Cosmet Laser Ther. 2014 Jan;16(1):32-6. doi: 10.3109/14764172.2013.854620. Epub 2013 Nov 19. PMID 24245880
- [Background] Bachmann F, Erdmann R, Hartmann V, Wiest L, Rzany B. The spectrum of adverse reactions after treatment with injectable fillers in the glabellar region: results from the Injectable Filler Safety Study. Dermatol Surg. 2009 Oct;35 Suppl 2:1629-34. doi: 10.1111/j.1524-4725.2009.01341.x. PMID 19807757
- [Background] Kassir R, Kolluru A, Kassir M. Extensive necrosis after injection of hyaluronic acid filler: case report and review of the literature. J Cosmet Dermatol. 2011 Sep;10(3):224-31. doi: 10.1111/j.1473-2165.2011.00562.x. PMID 21896135
- [Derived] Roh NK, Kim MJ, Lee YW, Choe YB, Ahn KJ. A Split-Face Study of the Effects of a Stabilized Hyaluronic Acid-Based Gel of Nonanimal Origin for Facial Skin Rejuvenation Using a Stamp-Type Multineedle Injector: A Randomized Clinical Trial. Plast Reconstr Surg. 2016 Mar;137(3):809-816. doi: 10.1097/01.prs.0000480686.68275.60. PMID 26910661

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Restylane Vital
Started | 25
Completed | 24
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Restylane Vital
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (8)
Age, Customized [Number; unit: participants]
  20-29 years | 4
  30-39 years | 14
  40-49 years | 5
  50-59 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 7
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 25
hydration [Mean (Standard Deviation); unit: AU (Arbitrary Unit)] — We measured a hydration level by a combination corneometer/mexameter/reviscometer device (Courage & Khazaka, Cologne, Germany).
  The range of hydration level was 0~120 AU(Arbitrary Unit).
  < 30 : Very dry, 30~49 : Dry, 50~59: Moisturized, >60 : Sufficiently Moisturized
  AU (Arbitrary Unit)
    treated side | 45.47 (10.53)
    untreated side | 46.21 (11.35)
elasticity [Mean (Standard Deviation); unit: AU (arbitrary unit)] — We measured a elasticity by a combination corneometer/mexameter/reviscometer device (Courage & Khazaka, Cologne, Germany).
  The range of elasticity is 0~400 AU(Arbitrary Unit). The lower revisometer values reflect higher elasticity.
  AU (arbitrary unit)
    treated side | 294.32 (90.25)
    untreated side | 272.70 (96.89)
melanin index [Mean (Standard Deviation); unit: AU(arbitrary unit)] — We measured a melanin index by a combination corneometer/mexameter/reviscometer device (Courage & Khazaka, Cologne, Germany).
  The range of melamin index is 0~999 AU(Arbitrary Unit).
  0~49: Phototype I (celtic type), 50~99 : Phototype II (Caucasian type), 100~149 : Phototype III (European mixed type), 150~199 : Phototype IV (Mediterranean type), 200~299 : Phototype V (Asian/Indian type), 300~999 : Phototype VI (Black skin type) (This is only an approach. It is recommend that each user should develop an own interpretation scale.)
  AU(arbitrary unit)
    treated side | 133.97 (25.56)
    untreated side | 133.66 (27.68)
erythema index [Mean (Standard Deviation); unit: AU(arbitrary unit)] — We measured a erythema index by a combination corneometer/mexameter/reviscometer device (Courage & Khazaka, Cologne, Germany).
  The range of erythema index is 0~999 AU(Arbitrary Unit). The lower erythema indices than baseline reflect improvement of erythema.
  AU(arbitrary unit)
    treated side | 292.74 (71.64)
    untreated side | 290.50 (59.35)

OUTCOME MEASURES:

1. Primary Outcome: Hydration Level
Description: We measured a hydration level by a corneometer device (Courage & Khazaka, Cologne, Germany).
  The range of hydration level was 0 (as dry as possible) ~120 AU (Arbitrary Unit)(most moist possible)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: AU (arbitrary unit)
Groups:
- Treated Side (Restylane Vital): stabilized hyaluronic acid (HA)-based gel of nonanimal origin
  Restylane Vital: stabilized hyaluronic acid (HA)-based gel of nonanimal origin
- Untreated Side: Eligible patients received injections of NASHA into the dermis on one side of the lower part of the cheek in a single session, at the start of the study (visit 1); the other side was left untreated.
Arm/Group | Treated Side (Restylane Vital) | Untreated Side
Number analyzed (Participants) | 24 | 24
AU (arbitrary unit) | 53.19 (9.08) | 46.75 (9.24)
Statistical Analysis 1: Comparison: Treated Side (Restylane Vital) vs Untreated Side; The change in each of the biophysical parameters was calculated as the pretreatment value minus the posttreatment value for each visit, and these pre- vs posttreatment changes were used in the statistical analysis to minimize the intraindividual variation between the two cheeks. The Wilcoxon rank-sum test was performed to compare the week-by-week changes in parameters of the right and left cheeks (i.e., treated vs untreated); Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Elasticity
Description: We measured a elasticity by a reviscometer device (Courage & Khazaka, Cologne, Germany).
  The range of elasticity was 0 (most elastic possible as) ~400 AU(Arbitrary Unit) (inelastic as possible)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: AU (arbitrary unit)
Arm/Group | Treated Side (Restylane Vital) | Untreated Side
Number analyzed (Participants) | 24 | 24
AU (arbitrary unit) | 242.33 (72.21) | 271.15 (86.10)
Statistical Analysis 1: Comparison: Treated Side (Restylane Vital) vs Untreated Side; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Melanin Index
Description: We measured a melanin index by a mexameter device (Courage & Khazaka, Cologne, Germany).
  The range of melanin index was 0 (as bright as possible) ~999 AU (Arbitrary Unit) (most dark possible).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: AU (arbitrary unit)
Arm/Group | Treated Side (Restylane Vital) | Untreated Side
Number analyzed (Participants) | 24 | 24
AU (arbitrary unit) | 147.25 (27.46) | 149.00 (26.86)
Statistical Analysis 1: Comparison: Treated Side (Restylane Vital) vs Untreated Side; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Erythema Index
Description: We measured an erythema index by a mexameter device (Courage & Khazaka, Cologne, Germany).
  The range of erythema index is 0~999 AU(Arbitrary Unit). The range of erythema index was 0 (as non-erythematous as possible) ~999 AU (most erythematous possible)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: AU (arbitrary unit)
Arm/Group | Treated Side (Restylane Vital) | Untreated Side
Number analyzed (Participants) | 24 | 24
AU (arbitrary unit) | 253.66 (58.19) | 243.53 (51.65)
Statistical Analysis 1: Comparison: Treated Side (Restylane Vital) vs Untreated Side; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Global Aesthetic Improvement Scale (Investigator)
Description: The therapeutic outcome was assessed by investigator using the Global Aesthetic Improvement Scale (GAIS), which rates outcome on the following 5-point scale: 3, very much improved; 2, much improved; 1, improved; 0, no change; and -1, worse.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Treated Side (Restylane Vital) | Untreated Side
Number analyzed (Participants) | 24 | 24
scores on a scale | 1.38 (0.77) | 0 (0)
Statistical Analysis 1: Comparison: Treated Side (Restylane Vital); The therapeutic outcome was assessed by patient self-assessment using the Global Aesthetic Improvement Scale, which rates outcome on the following 5-point scale: 3, very much improved; 2, much improved; 1, improved; 0, no change; and -1, worse. Two independent investigators also individually assessed every patient's improvement, and the values of the two scores were averaged for each patient. The Wilcoxon rank-sum test was performed to compare the pre-by-posttreatment changes in treated side; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Global Aesthetic Improvement Scale (Subject)
Description: The therapeutic outcome was assessed by patient self-assessment using the Global Aesthetic Improvement Scale (GAIS), which rates outcome on the following 5-point scale: 3, very much improved; 2, much improved; 1, improved; 0, no change; and -1, worse
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Treated Side (Restylane Vital) | Untreated Side
Number analyzed (Participants) | 24 | 24
scores on a scale | 1.33 (1.05) | 0 (0)
Statistical Analysis 1: Comparison: Treated Side (Restylane Vital); [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 12weeks
Description: Adverse events were self-reported by the patients completing a questionnaire.
Arm/Group | Restylane Vital
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 24/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restylane Vital (N=24)
erythema (Skin and subcutaneous tissue disorders) | 24 (24) — Erythema developed right after the treatment and maintained until 5days after the treatment

LIMITATIONS AND CAVEATS:
First, it did not have a double-blind design, and so the GAIS scores of the subjects could have been influenced. Second, the posttreatment follow-up period was relatively short, at 12 weeks. Finally, the patient sample in this study was small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No